CLINICAL TRIAL: NCT05808088
Title: The Effect of Hypnotherapeutic Sound-files on the Sleep of Parents in the Neonatal Unit.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HGO1
Record Dates: First submitted 2023-03-16; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Parents; Sleep; Infant, Premature; Hypnosis
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: One group receives the intervention at inclusion, the other group is a control group, but crosses over to intervention halfway through the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1, sound-files from inclusion (Experimental)
  Interventions: Other: Hypnotherapeutic sound-files
- Group 2, sound-files after 7 days (Active Comparator)
  Interventions: Other: Hypnotherapeutic sound-files

INTERVENTIONS:
Other: Hypnotherapeutic sound-files — The participants have access to hypnotherapeutic sound files which they can use as the please.

SUMMARY:
The goal of this randomised study is to learn about, the effect of hypnotherapeutic sound-files on the sleep of parents of infants in the neonatal unit. The main questions it aims to answer are:

* Can hypnotherapeutic sound-files make parents of infants in the neonatal unit sleep longer and better?
* Does hypnotherapeutic sound-files effect the state anxiety score of parents of infants in the neonatal unit?

Participants will have access to sound-files and:

* wear actigraphy sleep registration
* complete state-trait anxiety score

ELIGIBILITY:
Inclusion Criteria:

* Parents of a newborn in the neonatal unit at Randers Regional Hospital

Exclusion Criteria:

* Age under 18
* Hearing disability to an extend where sound-files cannot be used
* Psychotic diagnosis, including schizophrenia and personality disorder
* Already using hypnotherapeutic sound-files
* The use of sleep medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Sleep duration | Actigraphy will be worn 2 weeks
  Via actigraphy sleep duration is measured in minutes
Sleep quality | Actigraphy will be worn 2 weeks
  Sleep quality is data from actigraphy

SECONDARY OUTCOMES:
State Anxiety | State Anxiety score are measured at Baseline ( inclusion), day 7 and day 14
  State-Trait Anxiety Score
Trait Anxiety | Trait Anxiety Score are measured at Baseline (inclusion).
  State-Trait Anxiety Score

CONTACTS AND LOCATIONS:
Overall Officials: Helle Olesen, Principal Investigator — Randers Regional Hospital
Locations (1):
- Randers Regional Hospital, Randers, Denmark

IPD SHARING:
Plan to Share IPD: No